CLINICAL TRIAL: NCT03031236
Title: Effect of Integrated Management of Childhood Maltreatment, Maternal Depression, Psychosocial Stimulation and Nutritional Intervention on Child Development - A Randomized Controlled Trial
Brief Title: Reduce Childhood Maltreatment and Promote Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: UBS Optimus Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR-15002
Record Dates: First submitted 2016-11-13; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: Maltreatment
Keywords: Early Childhood Development (ECD); Psychosocial stimulation; Cognition; Parenting; Malnutrition; Bangladesh; Childhood Maltreatment
MeSH Terms: conditions — Malnutrition | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECD+ (Active Comparator): Behavioral: Psychosocial stimulation, Cognitive behavioral therapy and positive parenting practice The mothers of intervention (ECD+HN) group will receive fortnightly group sessions for 12 months that will include combined messages on a) psychosocial stimulation, b) positive parenting to prevent child maltreatment and c) cognitive behavioural therapy (CBT) for positive thinking, d) health and nutrition messages and e) 15 micronutrient sprinkle supplement.(90 sachets of over 6 month-period)
  Interventions: Behavioral: Psychosocial stimulation, Cognitive behavioral therapy and positive parenting practice
- Only regular health messages (No Intervention): Only regular health message from government health services

INTERVENTIONS:
Behavioral: Psychosocial stimulation, Cognitive behavioral therapy and positive parenting practice — The mothers of intervention (ECD+HN) group will receive fortnightly group sessions for 12 months that will include combined messages on a) psychosocial stimulation, b) positive parenting to prevent child maltreatment and c) cognitive behavioural therapy (CBT) for positive thinking, d) health and nutrition messages and e) 15 micronutrient sprinkle supplement.(90 sachets of over 6 month-period)
  Arms: ECD+

SUMMARY:
Background (brief):

1. Burden: The uniqueness of each child is tremendously influenced by interaction between nature and nurture during critical period of brain development that promotes foundation of brain architecture through neuronal connections.
2. Knowledge gap: Young children in Bangladesh are prone to multiple physiological and psycho-social risk factors e.g. poverty, maltreatment, malnutrition, disease, parental illiteracy, maternal depression and lack of stimulation, all of which are preventable. Little is reported about any comprehensive package of development that addresses most of these early childhood risks and promotes optimum early childhood development (ECD).
3. Relevance: The aim of this study is to develop and evaluate an integrated, low cost, and feasible center based approach that focuses on positive parenting of children during early life that will promote early stimulation, minimize childhood maltreatment, boost up of maternal self-esteem and healthy thinking and improve health and nutritional (HN) status of children.

Hypothesis (if any):

This integrated intervention will promote maternal child-care practices and mental health that will finally improve their children's growth, micro-nutrient status, early brain development compared to control group.

Objectives:

To see the effect of an integrated intervention (ECD + HN) on growth, micro-nutrient status, child development along with effect on maternal child-care practices and mental health.

Methods:

Randomly selected 2 groups will be identified as intervention and control (150 mothers' from15 clusters in each group). Mothers of 8-23 months old children living in slums and practice harsh child-disciplining will be identified as study population. The mothers of intervention (ECD+HN) group will receive fortnightly group sessions for 11 months that will include combined messages on a) psycho-social stimulation, b) positive parenting to prevent child maltreatment and c) cognitive behavioral therapy (CBT) for positive thinking, d) health and nutrition messages and e) 15 micro-nutrient sprinkle supplement.(90 sachets of over 6 month-period). The control group will only receive the usual health messages provided by the government.

Outcome measures/variables:

* Children's cognitive, motor, language and socio-emotional development; anthropometry; hemoglobin and micro-nutrient status (serum vitamin B12, iron and folic acid)
* Mother s' parenting practices, depressive symptoms, self-esteem and child-maltreatment.

DETAILED DESCRIPTION:
Hypothesis to be tested:

This integrated intervention will a) improve children's growth, hemoglobin, micro-nutrient status (vitamin B12 and folic acid), cognitive, motor, language and social-emotional development, b) minimize maltreatment of children by parents, c) improve positive parenting and d) reduce mothers' stress and depressive symptoms compared to control group.

Objectives:

Primary: This integrated intervention will

* Improve cognitive, motor, language and social-emotional development of children
* Minimize maltreatment of children by the caregivers

Secondary: This integrated intervention will bring following benefits in intervention group compared to control group- On children-

* Improve height, weight and head circumference
* Improve hemoglobin, vitamin B12 and folic acid status, On mothers (primary caregivers)
* Reduce mothers' stress and depressive symptoms
* Improve positive parenting practices

Background of the Project including Preliminary Observations:

The rate of global acute malnutrition is 16% while the rate of stunting in Bangladesh is as high as 41% in <five yrs children. Moreover, the children in Bangladesh are either deficient in different micro-nutrients like iron 10.7% and iodine 34% or have inadequate micro-nutrients in their diets like vitamin B12 and folate which is less than 50%. Many children in developing countries fail to reach their developmental potential due to lack of cognitive stimulation and Bangladeshi children have limited access to play materials and activities.

According to Walker and colleagues 300 million children are exposed to violence globally. Our unpublished data show that 32% of children <2 years are subjected to maltreatment and harsh punishment in Bangladesh.

Depression is one of the leading causes of disease burden for women and children of these mothers may suffer from behavioral problems.. Depression is reported as a leading cause of disease burden for women aged 15-44 years in all countries. The South Asia has the least woman-friendly societies in the world. Maternal depression is becoming a major public health problem in these societies, partly due to gender roles and practices and partly to poverty. Depression indicates state of mind that causes symptoms like crying spells, sleeping problems, depressed mood, irritability, fatigue, anxiety, poor concentration and interpersonal hypersensitivity, and these can range from mild to severe in nature. Maternal depression not only affects mothers' health, evidenced by poorer nutrition, higher suicide attempts and self harm but also results in poor health and developmental outcomes of their children.

In Bangladesh prevalence of anxiety and depressive symptoms are as high as 18-33% and we found a significant association with child maltreatment in an urban community on). Rahman et al. tested an innovative model of community-based management of depression using Cognitive Behavioral Therapy (CBT) in Pakistan and reported improvement in maternal depression 6 months postpartum. Considering similar family structure, religion and culture between Bangladesh and Pakistan, it is likely that the program will work in Bangladesh too.

Despite prevalent child maltreatment in Bangladesh, there are very few interventions to reduce maltreatment and those for children under 5 yrs of age are even rarer. Similarly, though attention has been diverted to ECD for several years now, very few of those programs address children under 3 yrs of age. Study design would probably be the 1st intervention using a robust research method to test the efficacy of an integrated method to address ECD, child maltreatment as well as health and nutrition of young children. Investigators will modify existing curriculum to further focus on child maltreatment. Investigators have targeted poor families from urban slums who are deprived of such services but face most of the risk factors and hope to improve their families' condition using low-cost intervention. Researchers have targeted the mothers as study participants who also primary caregiver of a child especially at younger age and have a major role in the child development. Mothers are also more vulnerable for depression than the fathers in Bangladeshi culture.

In addition, there is no culturally appropriate tool to assess child maltreatment in Bangladesh. In this project researchers attempt to modify or adapt existing instruments or if needed develop new tools suitable for use in Bangladesh.

Research Design and Methods

Population and sample size:

This study will be conducted in the semi-urban area (preferably in Kamalapur) of Dhaka, Bangladesh. Total sample is 10 mother-child duos in randomly selected 30 clusters ( n=300), half of which (n=150) will be beneficiaries from the intervention.

Plan of work: The intervention package will be piloted in the non study community for its feasibility and will be modified accordingly. The selected mother-child duos will be invited to field office for baseline assessments. Intervention group will be invited to join the center-based group sessions fortnightly for one year, the control group will receive existing government health messages. Both the groups will receive free health service from study medical officer for acute illnesses. After a year, final assessments will be done in both the groups. At baseline and end line mother-child interaction will be observed in a sub-sample of the population.

Procedures:

It will be a cluster-randomized trial. Clusters will be formed based on number of household members (those using the same cooking pot) as well as geographical boundary. On average there will be 150-200 households in each cluster, but there may be some variation in household numbers per cluster and per stratum.Total sample will be 10 mother-child duos in randomly selected 30 clusters (n=300), half of which (n=150) will be beneficiaries from the intervention.

Plan of work: The intervention package will be piloted in the non study community for its feasibility and will be modified accordingly. The selected mother-child duos will be invited to field office for baseline assessments. Intervention group will be invited to join the center-based group sessions fortnightly for 1 year, the control group will receive existing government health messages. Both the groups will receive free health service from study medical officer for acute illnesses. After a year, final assessments will be done in both the groups. At baseline and end line mother-child interaction will be observed in a sub-sample of the population. At the beginning of the study, 4 Focus group discussions of (8-10 non-study mothers) will be conducted in the community to know about the mothers' parenting practices. At the middle of the study qualitative information (case report and 30 In-Depth Interviews) will be collected form the intervened mothers about the intervention package they are receiving. Intervened mothers will be interviewed at their home according to their time availability. Key Informant's Interview (KII) will be conducted after a year from 2 play leaders (who will deliver the intervention) and 2 supervisors (who will train the play leaders and monitored them). Interviews will be taken and tape recorded with consent of the participants.

1. Preparatory works: At the first phase researchers will select the site and also complete the process of 'Ethical Review' of the project.

   Screening and enrollment: After taking the consent, screening of mothers of 8 to 23 months old children, who practice harsh discipline will be conducted in 30 identified clusters by trained health workers using ISPCAN Child Abuse Screening Tool-Parent Version (ICAST-P). Researchers have already used the modified version of these tools in Bangladesh. According to primary investigation there are 10% mothers having 8 to 23 months old children in study field site. With this estimation to get 10 eligible mothers from each cluster researcher group have to screen 100 mothers. Mothers who will fulfill the study enrollment criteria will be offered to join the study and will be invited to the test centers for baseline assessments.

   At the same time research group will start developing the study materials:

   For intervention: Development and piloting of following manuals, that already exist and needs further simplification and adaptations
   * Psycho-social stimulation for individual visits
   * Cognitive behavioral therapy For assessments: Cultural adaptation, Standard Operating Procedures (SOPs) preparation and field testing of following tools
   * Bayley Scale of Infant and Toddler Development (Already adapted, we have to take permission from Pearson's to use it)
   * Field testing and adaptation of ISPCAN Child Abuse Screening Tool -Parent Version (ICAST-P)
   * Qualitative questionnaires
   * Observational tools

   Tools that are adapted, tested and ready to use
   * Parenting questionnaire
   * Home observation for measurement of environment (HOME)
   * Rosenberg Self Esteem Scale
   * CES-D to measure depressive symptoms
   * Socio-economic status (SES) questionnaire
   * Wolke's Behavior Rating scale
   * Anthropometric measurements
2. Baseline assessment:

   On children:

   Bayley Scales of Infant and Toddler Development (Bayley-III) will be used to assess cognitive, language and motor development of the children. The test has been used in many developing countries, and has been the instrument of choice for much nutrition and child development research at this age in other countries like Indonesia and Brazil. The Bayley has often been sensitive to changes following interventions. Because the Bayley has not been standardized in Bangladesh, researcher will not compare these children's scores with the test norms or children of other countries. Study aim is only to compare the development of groups of children within the same community. Bayley usually takes about an hour to test the children.

   The children's behavior during the Bayley tests will be rated on five 9-point scales using a modified version of the scales developed by Wolke (1990). These ratings include infants' activity (very still=1 to overactive=9), emotional tone (unhappy=1 to radiates happiness=9), approach or responsiveness to examiner in the first 10 minutes (avoiding=1to friendly and inviting=9), cooperation with test procedure (resists all suggestions=1to always complies=9), and vocalization (very quiet=1to constant vocalization=9). The scale has been used in several studies in Bangladesh and was sensitive to intervention effects .

   Anthropometry: Mother and child's anthropometric measurements (height and weight of mothers; length/height, weight, MUAC and head circumference of children) will be assessed at using standard procedures.

   On mothers':

   Maternal self esteem: This will be assessed using adapted version of the Rosenberg Self Esteem Scale, the most widely used measure of self esteem for research purposes. It has been used previously in Bangladesh by this research team and by others as a valid instrument.

   Information on child maltreatment and neglect: The International Society for the Prevention of Child Abuse and Neglect (ISPCAN) has developed ISPCAN Child Abuse Screening Tool- Parent Version (ICAST-P) that has been widely used in developing countries, like India and Jamaica. This research group already used modified version of this tool in Bangladesh on hospital mothers.

   Measurement of maternal depressive symptoms will be done using Center for Epidemiologic Studies Depression Scale (CES-D). This tool has been used in Bangladesh and South-East Asian countries.

   Quality of stimulation at home was assessed using Caldwell's Home Observation for Measurement of Environment (HOME) which was modified for Bangladesh and was used in other studies by the same research team.

   Other measurements: These following measures will be collected as covariates - Socioeconomic status: On enrollment information will be collected on the family's assets (furniture e.g. bed/tables/chairs, electrical household equipment's e.g. radio/TV/fan, farm animals, vehicles e.g. rickshaw/boat/bicycle/motorbike, etc.), housing condition (type of roof, floor and walls), access to water and sanitation, electricity, crowding condition, and parental education and occupation. An asset quintile will be created from all available assets available at household level.

   Observational tools: Structured observation checklist will be used to see mother-child interaction Qualitative assessments will be used to conduct focus group discussion, in depth interviews and case reports.
3. Intervention:

It will be a low cost intervention focusing on building awareness among population at risk through hands on training delivered by trained health workers with minimum educational level and low salary. Our previous experience shows that it is possible to train paraprofessionals to provide intervention of this intensity. We have also shown that psycho-social stimulation provided for 10 or 12 months can improve the development and behavior of children significantly. Two weeks training and one week's field practice will be required to train these staff. We will train the play leaders regarding the whole intervention package including stimulation, Cognitive Behavioral Therapy, health and nutrition messages that include infant and young child feeding practices, good hygiene practice, and positive parenting messages (stimulation, learning through play, love and affection). There will be one-hour sessions fortnightly for 11 months. Attending 2 sessions per month is feasible for the mothers. This intervention will address the major risk factors e.g. negative parenting, lack of stimulation, child maltreatment, malnutrition, maternal stress/depressive symptoms, faulty care-seeking practices due to knowledge gap, etc. using a combined package.

There will be a combination of 3 types of interventions:

(i) Early stimulation and prevention of maltreatment through positive parenting, boosting up of maternal self-esteem and stress management (ECD): Psycho-social stimulation intervention will follow a set of culturally appropriate, semi-structured, child's age appropriate curriculum. This integrated approach will be given in groups of mothers and child. During the session the field-workers will show the mothers how to play with home-made toys and books and interact with their children in a way to promote their development. Along with the stimulation program, the field workers will also provide some advice regarding positive parenting and boosting up maternal self esteem and stress management. Care will be taken to appreciate mothers for their activities and positive reinforcement will be strongly encouraged. The developmental activities will be conducted in a playful manner and not as a work-oriented activity. The activities in the curriculum will be ordered by difficulty level and the health workers will be trained to choose the level for each child according to their ability to do the activities.

(ii) Health education and sprinkles supplementation (HN): The participants will receive health and nutrition messages to improve children's health. In addition children will receive multiple micro-nutrient powder (Vitamin A 400 µg, vitamin D 5 µg, vitamin E 5 mg, vitamin C 30 mg, thiamine 0.5 mg, riboflavin 0.5 mg, niacin 6 mg, pyridoxine 0.5 mg, vitamin B12 0.9 mg, folate 150 µg, iron 10 mg, zinc 4.1 mg, copper 0.56 mg, selenium 17.0 µg and iodine 90 µg) supplementation at household level (90 sachets of over 6 month-period).

(iii) Cognitive Behavioral Therapy: Intervention to help mothers change their negative behaviour and to improve self care, child care, income generation activities, will follow the "Thinking Healthy Program" model of Rahman and colleague using cognitive behavior therapy (CBT). CBT will improve maternal behaviour leading to "positive parenting" and prevention of maltreatment. Cognitive Behavioral Therapy is an "evidence-based and structured form of talking therapy that aims to alter the cycle of unhelpful or unhealthy thinking (cognition) and the resulting undesirable actions (behavior)." Cognitive Behavioral Therapy specifically focused on "changing thinking style toward positive" and not associated with any medication. CBT found to be effective in managing or treating not only depression, also a variety of other conditions-e.g. mood, personality, stress, eating habit, tic etc.This approach with rural mothers of similar context showed positive impact on child outcome in Pakistan, which is culturally and economically similar to Bangladesh.

CBT is aimed to alter the cycle of negative thinking of people to positive direction. The cycle of negative thoughts usually breaks in two ways by using Cognitive and Behavioral aspect of the therapy -

* Cognitive aspect of CBT: This focuses on altering ways of thinking of a person (mother) that includes thoughts, beliefs, ideas, attitudes, assumptions, mental imagery, and ways of directing her attention.
* Behavioral aspect of CBT: This focuses on helping the mother to face the challenges and the opportunities that facilitates child-raising with a sound and clear mind- and then to take necessary actions that are likely to have desired outcomes.

This model is proven to be an effective approach in breaking the cycle of depression and improving confidence, coping strategies and assertiveness in poor community with low resource setting. The cycle is broken through two ways of CBT- cognitive aspect (directing attention to positive direction) and behavioral aspect (helping to meet challenges).

d) Final assessment, data entry and data analysis: After 11 months of intervention, the participants will be invited again in the centre for end line assessment. The same assessment tools will be used as in the base line. Simultaneous data entry will continue in SPSS software. After data cleaning, preliminary analysis will be done according to following plan.

All the baseline variables will be used to compare between lost and tested groups as well as the intervention and control groups. The two time-point assessment will also provide information about within group changes. Some variables e.g. HOME, mother-child interaction, parenting, childcare etc. will be used either as mediator or as outcome in separate analyses

Outcome Variables:

On Mothers-

1. Maternal stress and depressive symptoms using CES-D at baseline and at the end.
2. Self Esteem assessment using Rosenberg Self Esteem Scale at baseline and at the end in test centre
3. Information about child maltreatment by parents will be collected at baseline during screening at home and at the end.
4. Home observation for measurement of environment (HOME) at household level, twice (at baseline and at the end)

On Children-

1. Child's cognitive, motor and language assessment using Bayley-III and behavioral assessment during test using Wolke's Behavior Rating Scale, at baseline and at the end in test centre. Children will accompany their mothers to the centre. (45 min)
2. Children's Micronutrient status (vitamin B12 and folic acid) at baseline and at the end in test centre
3. Children's Hemoglobin status
4. Children's height, weight, MUAC, head circumference at baseline and at the end

Covariates-

1. Socio-economic variables (asset index/ quintile)
2. Demographic variables (housing/ sanitation)
3. Maternal nutritional status (BMI)
4. Child's age and sex
5. Compliance on micro-nutrients and dietary recall
6. Morbidity Sample Size Calculation and Outcome (Primary and Secondary) Variable(s)

Considering 5% level of significance, 80% power, an improvement of 0.4 SD in children's developmental outcome based on our previous experiences, an ICC of 0.01 and 30% drop outs, we need to enroll 150 mother-child duos in each group as per equation below- 2(SD)2 n = ---------------- X f (αβ) (M1-M2) 2

n: sample required, SD: 16 (based on previous data of Bayley Score) α: 5% level of significance β: 80% power f= α*β M1-M2 = Difference = 6.4 points (based on previous studies) So the calculated n=100

Considering the clustering we need to adjust this sample size by multiplying the above value (100) by the design effect.

Design Effect = 1 + [(m-1) * ICC m corresponds to the average number of infants per cluster. Assuming there are on average 10 mother-child duos/cluster.

Using ICC = 0.01, the design effect = 1 + [(10-1) * ICC = 1 + 0.9 = 1.09 Therefore new sample size = 100*1.09= 109 per group , considering 30% drop-out the sample size per group is around 150 infants in stimulation group and 150 infants in control group.

Data Analysis

icddr,b scientists and co-investigators of this research project will analyze the data using Stata/SPSS. All data will be checked for normality. Log transformation will be done if not normally distributed. Indices will be created where it is required (eg: SES index, housing index etc). Pearson's correlations will be conducted to examine the association between age of the child and each developmental measure. A comparison will be done between the socio-demographic characteristics of the intervened and control groups using t-test for continuous variables and χ2 for categorical variables. Partial correlation will be used controlling age and sex to examine association of different covariates with developmental scores.

Finally, multi-level regression analyses will be done. In each regression analysis, the outcome will be the final developmental score, with age at enrollment, the relevant initial scores, and intervention as predictors. Again, comparison will be done between the treatment effect in intervention and control groups. All variables that will be different between intervention and control groups at baseline and will correlate with the developmental outcomes and will address high co-linearity among the covariates in all analyses.

The main outcomes are children's cognitive, language and motor development measured on Bayley Scales of Infant and Toddler Development. In addition it is expected that an improvement in growth, home stimulation and mother's positive parenting. It is also expected that improvement of the hemoglobin and micro-nutrient status (vitamin B12 and folic acid) over 150 children in the intervention group by the end of the project. At the same time it is expected of a reduction on mothers' stress and depressive symptom and rate of maltreatment of children by parents. A cost analysis will be conducted based on the success indicators, cost per successful outcome will be calculated from total cost of intervention program.

Data Safety Monitoring Plan (DSMP)

Researcher group do not expect the low risk activities of this study to put the study population at increased risk of adverse outcomes, however any human activity can have unforeseen untoward consequences. researchers will actively monitor the impact of the intervention on the population. The primary objective of these evaluations is to understand practices, knowledge, and attitudes towards the interventions. researchers will include questions in the evaluations that ask if they have noted any adverse outcomes.

If the field team learns of any adverse outcomes they will be trained to report them to the study team the same day they learn of them.

Ethical Assurance for Protection of Human rights

The project will have to be approved by the Institutional Review Board of icddr,b. Investigator group will collect written informed consent in Bengali from the parents before starting data collection. Research group will ensure confidentiality when collecting data on sensitive issues like maternal depression. Hard copies of the data will be kept in a locked cabinet only accessible to the investigators. The electronic data will not have the name and other identifiable information. Clinically depressed mothers will be referred to counsellors or psychiatrists as needed. Children with mental retardation or developmental disabilities will be referred to proper places for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of 8 to 23 months old children, who practice maltreatment or harsh child-discipline (screened by a previously used tool), will be included.
* Children 8-23 months old with weight-for-length ≥-3 z score, MUAC ≥ 115 mm
* Mothers are the primary caregivers and consented to participate.

Exclusion Criteria:

* severe malnutrition nutritional edema, known developmental disability, chronic illness, haemoglobin level <8 gm/L (at enrolment). They will be referred to the nearby health facilities for necessary clinical management

Ages: 8 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cognitive development (composite score of cognitive,motor, language and social-emotional development of children) | Change from baseline at 11 months of intervention
  cognitive development will be measured by Bayley tools. All individuals score will be aggregated in to composite score of cognitive,motor, language and social-emotional development of children

SECONDARY OUTCOMES:
Maltreatment of children by the caregivers | Change from baseline at 11 months of intervention
  The International Society for the Prevention of Child Abuse and Neglect (ISPCAN) has developed ISPCAN Child Abuse Screening Tool- Parent Version (ICAST-P) will be used for measuring the severity of maltreatment calculating score.
Height | Change from baseline at 11 months of intervention
  Height will be measure in centimeter through World Health Organization (WHO) guideline.
Weight | Change from baseline at 11 months of intervention
  Weight will be measure in gram through World Health Organization (WHO) guideline.
Head circumference | Change from baseline at 11 months of intervention
  Head circumference will be measure in centimeter through World Health Organization (WHO) guideline.
Haemoglobin | Change from baseline at 11 months of intervention
  The Hematological measurement will be measured as Hb per g/dl ,
vitamin B12 | Change from baseline at 11 months of intervention
  vitamin B12 will be measured as Pg/ml
folic acid status | Change from baseline at 11 months of intervention
  folic acid status will be measured as ng/ml
Retinol | Change from baseline at 11 months of intervention
  The Hematological measurement will be measured as Retinol per Mg /ml
STfR per Mg/ml | Change from baseline at 11 months of intervention
  The Hematological measurement will be measured as STfR per Mg/ml
Mothers' stress and depressive symptoms | Change from baseline at 11 months of intervention
  the Rosenberg Self Esteem Scale (Rosenberg, 1965), the most widely used measure of self esteem for research purposes and Measurement of maternal depressive symptoms will be done using Center for Epidemiologic Studies Depression Scale (CESD)
Positive parenting practices, | Change from baseline at 11 months of intervention
  A questionnaire will be used to measure positive parenting

CONTACTS AND LOCATIONS:
Overall Officials: Fahmida Tofail, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Fahmida Tofail, PhD, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black MM, Baqui AH, Zaman K, El Arifeen S, Black RE. Maternal depressive symptoms and infant growth in rural Bangladesh. Am J Clin Nutr. 2009 Mar;89(3):951S-957S. doi: 10.3945/ajcn.2008.26692E. Epub 2009 Jan 28. PMID 19176729
- [Background] Black MM, Baqui AH, Zaman K, McNary SW, Le K, Arifeen SE, Hamadani JD, Parveen M, Yunus M, Black RE. Depressive symptoms among rural Bangladeshi mothers: implications for infant development. J Child Psychol Psychiatry. 2007 Aug;48(8):764-72. doi: 10.1111/j.1469-7610.2007.01752.x. PMID 17683448
- [Background] Arsenault JE, Yakes EA, Islam MM, Hossain MB, Ahmed T, Hotz C, Lewis B, Rahman AS, Jamil KM, Brown KH. Very low adequacy of micronutrient intakes by young children and women in rural Bangladesh is primarily explained by low food intake and limited diversity. J Nutr. 2013 Feb;143(2):197-203. doi: 10.3945/jn.112.169524. Epub 2012 Dec 19. PMID 23256144
- [Background] Beck CT. Maternal depression and child behaviour problems: a meta-analysis. J Adv Nurs. 1999 Mar;29(3):623-9. doi: 10.1046/j.1365-2648.1999.00943.x. PMID 10210459
- [Background] Caldwell BM. Descriptive evaluations of child development and of developmental settings. Pediatrics. 1967 Jul;40(1):46-54. No abstract available. PMID 6028898
- [Background] Grantham-McGregor S; International Child Development Committee. Early child development in developing countries. Lancet. 2007 Mar 10;369(9564):824. doi: 10.1016/S0140-6736(07)60404-8. No abstract available. PMID 17350449
- [Background] Grantham-McGregor SM, Lira PI, Ashworth A, Morris SS, Assuncao AM. The development of low birth weight term infants and the effects of the environment in northeast Brazil. J Pediatr. 1998 Apr;132(4):661-6. doi: 10.1016/s0022-3476(98)70357-9. PMID 9580767
- [Background] Hamadani JD, Fuchs GJ, Osendarp SJ, Khatun F, Huda SN, Grantham-McGregor SM. Randomized controlled trial of the effect of zinc supplementation on the mental development of Bangladeshi infants. Am J Clin Nutr. 2001 Sep;74(3):381-6. doi: 10.1093/ajcn/74.3.381. PMID 11522564
- [Background] Hamadani JD, Fuchs GJ, Osendarp SJ, Huda SN, Grantham-McGregor SM. Zinc supplementation during pregnancy and effects on mental development and behaviour of infants: a follow-up study. Lancet. 2002 Jul 27;360(9329):290-4. doi: 10.1016/S0140-6736(02)09551-X. PMID 12147372
- [Background] Hamadani JD, Huda SN, Khatun F, Grantham-McGregor SM. Psychosocial stimulation improves the development of undernourished children in rural Bangladesh. J Nutr. 2006 Oct;136(10):2645-52. doi: 10.1093/jn/136.10.2645. PMID 16988140
- [Background] Walker SP, Wachs TD, Grantham-McGregor S, Black MM, Nelson CA, Huffman SL, Baker-Henningham H, Chang SM, Hamadani JD, Lozoff B, Gardner JM, Powell CA, Rahman A, Richter L. Inequality in early childhood: risk and protective factors for early child development. Lancet. 2011 Oct 8;378(9799):1325-38. doi: 10.1016/S0140-6736(11)60555-2. Epub 2011 Sep 22. PMID 21944375
- [Background] Idjradinata P, Pollitt E. Reversal of developmental delays in iron-deficient anaemic infants treated with iron. Lancet. 1993 Jan 2;341(8836):1-4. doi: 10.1016/0140-6736(93)92477-b. PMID 7678046
- [Background] Karasz A. Cultural differences in conceptual models of depression. Soc Sci Med. 2005 Apr;60(7):1625-35. doi: 10.1016/j.socscimed.2004.08.011. PMID 15652693
- [Background] Khan MM, Reza H. The pattern of suicide in Pakistan. Crisis. 2000;21(1):31-5. doi: 10.1027//0227-5910.21.1.31. PMID 10793469
- [Background] Kumar V. Poisoning deaths in married women. J Clin Forensic Med. 2004 Feb;11(1):2-5. doi: 10.1016/j.jcfm.2003.10.010. PMID 15261005
- [Background] Lawrence V, Murray J, Banerjee S, Turner S, Sangha K, Byng R, Bhugra D, Huxley P, Tylee A, Macdonald A. Concepts and causation of depression: a cross-cultural study of the beliefs of older adults. Gerontologist. 2006 Feb;46(1):23-32. doi: 10.1093/geront/46.1.23. PMID 16452281
- [Background] Lind T, Lonnerdal B, Stenlund H, Gamayanti IL, Ismail D, Seswandhana R, Persson LA. A community-based randomized controlled trial of iron and zinc supplementation in Indonesian infants: effects on growth and development. Am J Clin Nutr. 2004 Sep;80(3):729-36. doi: 10.1093/ajcn/80.3.729. PMID 15321815
- [Background] Lovejoy MC, Graczyk PA, O'Hare E, Neuman G. Maternal depression and parenting behavior: a meta-analytic review. Clin Psychol Rev. 2000 Aug;20(5):561-92. doi: 10.1016/s0272-7358(98)00100-7. PMID 10860167
- [Background] Murray L, Cooper P. Effects of postnatal depression on infant development. Arch Dis Child. 1997 Aug;77(2):99-101. doi: 10.1136/adc.77.2.99. No abstract available. PMID 9301345
- [Background] Nasreen HE, Kabir ZN, Forsell Y, Edhborg M. Impact of maternal depressive symptoms and infant temperament on early infant growth and motor development: results from a population based study in Bangladesh. J Affect Disord. 2013 Apr 5;146(2):254-61. doi: 10.1016/j.jad.2012.09.013. Epub 2012 Oct 11. PMID 23063237
- [Background] Patel V, Rahman A, Jacob KS, Hughes M. Effect of maternal mental health on infant growth in low income countries: new evidence from South Asia. BMJ. 2004 Apr 3;328(7443):820-3. doi: 10.1136/bmj.328.7443.820. PMID 15070641
- [Background] Pollitt E, Saco-Pollitt C, Jahari A, Husaini MA, Huang J. Effects of an energy and micronutrient supplement on mental development and behavior under natural conditions in undernourished children in Indonesia. Eur J Clin Nutr. 2000 May;54 Suppl 2:S80-90. doi: 10.1038/sj.ejcn.1601009. PMID 10902991
- [Background] Raj A, Silverman JG. Intimate partner violence against South Asian women in greater Boston. J Am Med Womens Assoc (1972). 2002 Spring;57(2):111-4. PMID 11991419
- [Background] Schellenberg JA, Victora CG, Mushi A, de Savigny D, Schellenberg D, Mshinda H, Bryce J; Tanzania Integrated Management of Childhood Illness MCE Baseline Household Survey Study Group. Inequities among the very poor: health care for children in rural southern Tanzania. Lancet. 2003 Feb 15;361(9357):561-6. doi: 10.1016/S0140-6736(03)12515-9. PMID 12598141
- [Background] Segre LS, Stasik SM, O'Hara MW, Arndt S. Listening visits: an evaluation of the effectiveness and acceptability of a home-based depression treatment. Psychother Res. 2010 Nov;20(6):712-21. doi: 10.1080/10503307.2010.518636. PMID 21154029
- [Background] Tofail F, Hamadani JD, Mehrin F, Ridout DA, Huda SN, Grantham-McGregor SM. Psychosocial stimulation benefits development in nonanemic children but not in anemic, iron-deficient children. J Nutr. 2013 Jun;143(6):885-93. doi: 10.3945/jn.112.160473. Epub 2013 Apr 24. PMID 23616511
- [Background] Tsutsumi A, Izutsu T, Akramul Islam MD, Amed JU, Nakahara S, Takagi F, Wakai S. Depressive status of leprosy patients in Bangladesh: association with self-perception of stigma. Lepr Rev. 2004 Mar;75(1):57-66. PMID 15072127
- See also: Uddin MK, Islam MT, Asaduzzaman M. Perceived Stress and Self-Esteem as Significant Predictors of Cigarette Smoking Behavior of Bangladeshi Male Adults. — https://www.academia.edu/4936041/Perceived_Stress_and_Self-Esteem_as_Significant_Predictors_of_Cigarette_Smoking_Behavior_of_Bangladeshi_Male_Adults